CLINICAL TRIAL: NCT03030157
Title: Prospective Randomized Phase II Trial: Single Instillation Versus Long-term Prophylactic Intravesical Instillation of Pirarubicin in the Prevention of Bladder Recurrence After Nephroureterectomy for Primary Upper Tract Urothelial Carcinoma
Brief Title: Single Versus Long-term Intravesical Instillation Chemotherapy for Recurrence After Nephroureterectomy for Upper Tract Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pudong Hospital (Other); Shanghai Pudong New Area Gongli Hospital (Other)
Responsible Party: Principal Investigator, Yiran Huang, Director of Urology department in Renji Hospital, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RenJiH-PDU Trial
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Intravesical Instillation
Keywords: urothelial cancer; bladder cancer; nephroureterectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pirarubicin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long-term Intravesical Instillation of pirarubicin(THP) (Experimental): A single instillation of pirarubicin (THP) plus one year long-term intravesical instillation after nephroureterectomy was performed. The ﬁrst instillation was initiated within 72-168 hours after surgery, followed by four times weekly and 11 times monthly (16 times in total in one year time) . Every time, THP 30 mg in 30 mL of normal saline was delivered into the bladder through a catheter and was retained for 30 minutes.
  Interventions: Drug: pirarubicin(THP)
- Single Intravesical Instillation of pirarubicin (Active Comparator): A single intravesical instillation of THP after nephroureterectomy was performed. This instillation was initiated within 72-168 hours after surgery . THP 30 mg in 30 mL of normal saline was delivered into the bladder through a catheter and was retained for 30 minutes.
  Interventions: Drug: pirarubicin(THP)

INTERVENTIONS:
Drug: pirarubicin(THP)

SUMMARY:
Up to 30-40% of the patients may develop bladder recurrance after radical nephroureterectomy for primary upper tract urothelial carcinoma. Bladder tumor needs transurethral resection, which is associated with costs of treatment and potential poor prognosis. Although several randomized controlled trial have shown that prophylactic intravesical chemotherapy could prevent bladder tumor recurrence, the optimal schedule and duration of treatment are unkown. The investigators want to determine the efficiacy of single instillation versus long-term intravesical instillation of pirarubicin for bladder recurrence after radical nephrouretectomy for primary upper tract urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with upper tract urothelial carcinoma
* have no distant metastasis
* have an ECOG 0 to 2
* expected to receive radical nephroureterectomy

Exclusion Criteria:

* a prior history of bladder or synchronous bladder cancer
* administration of neoadjuvant chemotherapy
* the presence of severe complications
* deny to receive cytoscopy
* patients with advanced stage (T4)
* patients with contralateral UTUCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of bladder cancer in the first 12 month following nephroureterectomy | 12 month
  Bladder recurrence is judged on visual appearance, and histopathologic proof of recurrence was required.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 day, 1 month and 12 month
questionnaire for quality of life | baseline, 1 month and 12 month
  e.g QLQ C-30
progression-free survival | 12 month
  progression-free survival
cancer-specific survival | 12 month
  cancer-specific survival
overall survival | 12 month
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China